CLINICAL TRIAL: NCT00316537
Title: A Multicenter, Randomized Study of the Safety and Preliminary Efficacy of Low-Dose Nicotine Gel (ATG002) in Patients With Plantar Diabetic Foot Ulcers
Brief Title: Safety and Preliminary Efficacy Study of Nicotine Gel to Treat Diabetic Foot Ulcers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: CoMentis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATG002-121
Record Dates: First submitted 2006-04-17; First posted 2006-04-21 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Diabetic Foot Ulcers
Keywords: diabetes; foot ulcers; nicotine gel; wound healing
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — Drug Evaluation

INTERVENTIONS:
Drug: ATG002 (study drug)

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of low dose nicotine gel in patients with chronic diabetic ulcers

DETAILED DESCRIPTION:
This pilot study will be the first time that nicotine will be applied directly onto the surface of chronic diabetic ulcer. The goals of the study are to evaluate safety and tolerability (particularly at the wound site) of a gel formulation containing low-dose nicotine, and to obtain preliminary information on its effects on accelerating wound closure. The study will be carried out on a background of conventional wound therapy in patients with Type II diabetes mellitus. Patients will be randomized to receive either study medication (ATG002), vehicle gel, or standard-of-care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type II
* Single non-healing uninfected partial or full-thickness foot ulcer secondary to diabetic neuropathy, in the absence of significant peripheral arterial disease.

Exclusion Criteria:

* Patients who use tobacco in any form or who are on nicotine replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Assessment of ulcer size as determined by weekly ulcer tracings

SECONDARY OUTCOMES:
Assessment for complete wound closure. "Complete wound closure" will be defined as full epithelialization of the wound with the absence of drainage and lack of dressing requirement for an interval of at least 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Hsu, MD, Study Director — Athenagen, Inc.
Locations (13):
- United States (13):
  - SeniorCare, Alabama Geriatric Specialists, Homewood, Alabama
  - Hope Research Institute, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Center for Clinical Research, Castro Valley, California
  - University of San Diego Wound Treatment and Research Center, San Diego, California
  - University of Miami, Miami, Florida
  - Ankle and Foot Specialists of Atlanta, Lithonia, Georgia
  - Crossroads Research, Inc., Owings Mills, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - NewBridge Medical Research, Warren, Pennsylvania
  - Central Washington Podiatry Service, Yakima, Washington
  - Aurora Health Care / Lukes Medical Center, Milwaukee, Wisconsin